CLINICAL TRIAL: NCT04735094
Title: Randomized Control Trial of the Use and Effectiveness of Balloon for Endobronchial Ultrasonography.
Brief Title: The Use and Effectiveness of Balloon for Endobronchial Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT0101
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer Staging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endobronchial biopsy with the use of a balloon attached to the echo-bronchoscope (Experimental)
  Interventions: Diagnostic Test: Endobronchial biopsy with the use of a balloon attached to the echo-bronchoscope
- Endobronchial biopsy without the use of a balloon attached to the echo-bronchoscope (No Intervention)

INTERVENTIONS:
Diagnostic Test: Endobronchial biopsy with the use of a balloon attached to the echo-bronchoscope — A small balloon made of latex can be attached to the tip of echo-bronchoscope which is then inflated with water or saline for better apposition of the echo-endoscope and the airway wall. This may improve ultrasound image quality and aid better visualization of the lymph nodes.
  Arms: Endobronchial biopsy with the use of a balloon attached to the echo-bronchoscope

SUMMARY:
Although balloons appear to improve ultrasound image quality, it's use can be technically difficult for segmental airways because of anatomical limitations to convex probe imaging. Furthermore, it is uncertain whether this leads to a better diagnostic yield. To our knowledge, there are currently no studies showing that the use of balloon improves diagnostic yield with EBUS. We hypothesize that the use of balloon may increase the diagnostic yield by improving ultrasound image quality and reduce the duration of the procedure.The aim of this study is to analyse whether the use of balloon during linear EBUS 1) improves diagnostic yield, 2) reduces the duration of the procedure, and 3) improves ultrasound image quality with increased operator satisfaction in terms of ease of procedure.

ELIGIBILITY:
Inclusion criteria:

* Adults aged ≥18 years
* Patient referred for EBUS guided TBNA of mediastinal LNs
* The para-tracheal lymph node (LN) station 4R is planned to be biopsied.

Exclusion criteria

-Patient referred for EBUS and 4R is NOT planned to be biopsed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 1 year
  Diagnostic yield will be calculated separately for each group with and without the use of balloon. Diagnostic yield will be defined as a satisfactory sample with presence of lymphocytes in the aspirate on the final pathology report. In order to minimise the confounding factor in diagnostic yield based on the dimensions of the LN, we chose a single LN station (4R) and patients were sub-dvided into 3 groups based on the size of the LN.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided